CLINICAL TRIAL: NCT03109002
Title: Epidemiology of Treatment Resistant Depression in the US: Analysis of Health Services Databases
Brief Title: An Epidemiology Study of Treatment Resistant Depression in the United States (US)
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108308; RRA-18629 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-04-06; First posted 2017-04-11 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Treatment-Resistant
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Pharmacologically Treated Depression (PTD) Cases: This study is based on anonymized health services data, study population include US residents with medical insurance between 1 Jan, 2010 and 31 Dec, 2014 as described by the Truven MarketScan Medicaid (MDCD), Truven MarketScan Medicare Supplemental (MCDR), and Truven MarketScan Commercial Claims and Encounters (CCAE) databases. Within each database, pharmacologically treated depression (PTD) cases incident during 2011 will be followed for up to 4 years to ascertain their TRD status and 1-year incidence rates for PTD and TRD. Participants will not receive any intervention as a part of this study. To assure they are incident rather than prevalent cases, study participants are required to have 1 year without a dispensing of an antidepressant medication before they can join the cohort.

SUMMARY:
The purpose of this study is to describe the epidemiology of Treatment Resistant Depression (TRD) in the US, including the population incidence of TRD, and TRD as a proportion of Pharmacologically Treated Depression (PTD), and stratify the estimates by sex and age group, with separate estimates for the Medicaid population, the Medicare population, and the privately insured population. Anonymized participants data will be used for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Have been in the database for the past year (ignoring breaks of < 30 days)
* Have not had, an excluded diagnosis or dispensing of an AD medication during the past year
* Are aged 14 to 60 years (if in the CCAE or MCDC databases), or are aged greater than or equal to (>=) 65 years (if in the MCDR database). Age is defined as age on Jan 1, 2011. The boundary at age 60 for the first two databases is intended to avoid loss to follow-up due to transfer to Medicare at age 65. The boundary at age 65 for the MCDR database reflects the fact that very few people described by that database are aged less than 65

Exclusion Criteria:

- Participants will be excluded when they receive diagnoses Schizophrenia, Bipolar disorder including mania or Dementia

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: US residents with medical insurance between 1 Jan, 2010 and 31 Dec, 2014 will be assessed.
Sampling Method: Probability Sample
Enrollment: 200000 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2017-05-18 (Actual); Study Completion 2017-05-18 (Actual)

PRIMARY OUTCOMES:
Incidence Rate of Treatment Resistant Depression | Up to 4 years
  TRD will be defined as the failure of two medications, as marked by their replacement or supplementation with other medications using three alternative definitions. In one the time for a medication regimen to fail is limited to less than or equal to (<=) 3 months and in the second the time for a medication regimen to fail is limited to <= 6 months, both corresponding to the medication never providing adequate relief. In the third, the time for a medication regimen to fail will be limited to <= 2 years, corresponding to the medication not providing permanent or very long lasting relief.
Treatment Resistant Depression as a Proportion of Pharmacologically Treated Depression | Up to 4 years
  An episode of PTD begins when a member of the study cohort receives a dispensing of an antidepressant (AD) medication and receives a diagnosis of depression between 180 days before that dispensing and 30 days after that dispensing.
Incidence Rate of Treatment Resistant Depression by Age Group and Sex | Up to 4 years
  TRD incidence will be stratified by age group and sex under each of the three definitions of failure of a medication regimen.
Incidence Rate of TRD as Separate Estimates for the Medicaid Population, the Medicare Population, and the Privately Insured Population | Up to 4 years
  TRD incidence will be stratified by data population (database): Medicaid, Medicare, Privately insured.

SECONDARY OUTCOMES:
Incidence on TRD Based on Sensitivity Analysis | Up to 4 years
  Sensitivity analyses are intended to clarify how the results of the present study will compare to the results of other studies that may define as The maximum time for failure of a regimen is changed to: 60, 120, 150, or 365 days, or is not limited; the requirement that a regimen include greater than or equal to (>=) 28 days' supply of the antidepressant medication and antipsychotic medication (if present) is changed to >= 42 days and 14 days supply; participants who get an excluded diagnosis are retroactively excluded from the study cohort; or the definition of an incident case adds a requirement for no depression diagnosis in the prior year.
Number of Participants With Selected Markers for Severity of Depression | Up to 4 years
  The following markers of severity will be tabulated during the PTD episodes and stratified according to whether the participant develops or does not develop TRD during the study period: Electro-convulsive therapy, hospitalization with a diagnosis of depression, receiving a diagnosis of suicidal thoughts, receiving a diagnosis of self-harm, emergency department visit with a diagnosis of injury, emergency department visit with a diagnosis of poisoning.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC

IPD SHARING:
Plan to Share IPD: No
The data for this study came from health services databases to which access is available under contracts that limit further distribution.

REFERENCES:
- [Result] Fife D, Reps J, Cepeda MS, Stang P, Blacketer M, Singh J. Treatment resistant depression incidence estimates from studies of health insurance databases depend strongly on the details of the operating definition. Heliyon. 2018 Jul 26;4(7):e00707. doi: 10.1016/j.heliyon.2018.e00707. eCollection 2018 Jul. Erratum In: Heliyon. 2019 Mar 07;5(3):e01198. doi: 10.1016/j.heliyon.2019.e01198. PMID 30094377